CLINICAL TRIAL: NCT06275204
Title: Multicentric Transnational H. Pylori Screen-and-treat Study in a Population of Young Adults
Brief Title: H. Pylori Screen-and-treat Study in a Population of Young Adults
Status: Recruiting | Type: Observational
Sponsor: University of Latvia (Other)
Collaborators: Clinical Hospital Center Rijeka (Other); Clinical Hospital Centre Zagreb (Other); Beacon Hospital (Other); Wroclaw Medical University (Other); Iuliu Hatieganu University of Medicine and Pharmacy (Other); National Institute of Public Health, Slovenia (Other Government)
Responsible Party: Sponsor
Other Study IDs: 101101252; 101101252 (Other Grant/Funding Number: EU4H-2022-PJ-01)
Record Dates: First submitted 2024-02-08; First posted 2024-02-23 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer; H Pylori Infection; H Pylori Eradication; H-pylori
Keywords: H. pylori; gastric cancer; eradication therapy; screening
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Protocol I: H. pylori positive patients who will be treated by bismuth-based quadruple therapy.
  Participating centers: KBC Rijeka, Croatia; KBC Zagreb, Croatia; Beacon Hospital, Ireland; Uniwersytet medyczny we Wrocławiu, Poland; UMF Cluj-Napoca, Romania; NIJZ, Slovenia
  Interventions: Drug: Bismuth-based quadruple therapy
- Protocol II: In case there will be a treatment failure after bismuth-based quadruple therapy, the remaining patients with a positive infection will be referred to a levofloxacin based quadruple therapy.
  Participating centers: KBC Rijeka, Croatia; KBC Zagreb, Croatia; Beacon Hospital, Ireland; Uniwersytet medyczny we Wrocławiu, Poland; UMF Cluj-Napoca, Romania; NIJZ, Slovenia
  Interventions: Drug: Levofloxacin-based quadruple therapy
- Standard triple therapy: H. pylori positive participants who will offered standard triple therapy.
  Participating center: University of Latvia, Latvia
  Interventions: Drug: Standard triple therapy
- Second line treatment - levofloxacin-based: In case there will be a treatment failure after standart triple therapy, the remaining patients with a positive infection will be referred to a second line treatment
  Participating center: University of Latvia, Latvia
  Interventions: Drug: Levofloxacin-based triple

INTERVENTIONS:
Drug: Bismuth-based quadruple therapy — Participants who are positive with H. pylori will receive bismuth-based quadruple therapy:
  Antibiotic 1 - Amoxicillin 4 x 500 mg or Clarithromycin 2 x 400 mg, Antibiotic 2 - Metronidazole 4 x 400 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg, Colloidal bismuth - Bismuth oxide 4 x 120 mg.
  Groups: Protocol I
Drug: Levofloxacin-based quadruple therapy — In case there will be a treatment failure after Protocol I is completed, the remaining patients with a positive infection will be referred to a secondary treatment:
  Antibiotic 1 - Levofloxacin 1 x 500 mg, Antibiotic 2 - Metronidazole 4 x 400 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg, Colloidal bismuth - Bismuth oxide 4 x 120 mg.
  Groups: Protocol II
Drug: Standard triple therapy — Participants who are positive for H. pylori will receive a standard triple therapy:
  Antibiotic 1 - Amoxicillin 2 x 1000 mg, Antibiotic 2 - Clarithromycin 2 x 500 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg.
  Groups: Standard triple therapy
Drug: Levofloxacin-based triple — Participants with treatment failure will be recommended second line treatment - levofloxacin-based:
  Antibiotic 1 - Levofloxacin 2 x 500 mg, Antibiotic 2 - Amoxicillin 2 x 1000 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg
  Groups: Second line treatment - levofloxacin-based

SUMMARY:
Gastric cancer remains a major challenge to public health on a global scale. H. pylori related cancer burden contributes to the largest proportion of cancer cases attributable to infections in Europe. Considering its absolute burden and persisting disparities, in addition to the substantial prevalence of H. pylori infection worldwide that is treatable, gastric cancer is a logical target for urgent action for prevention. Population-based H. pylori test-and-treat has therefore been proposed as a strategy for gastric cancer prevention. To fill the gaps in knowledge about gastric cancer prevention through H. pylori screening and eradication in younger adults, a study of a population-based H. pylori test-and-treat strategy in Ireland, Croatia, Latvia, Poland, Romania and Slovenia.

Main goals of this study are to assess future program processes, feasibility, acceptability and effectiveness. In total of 6,800 adults aged 30-34 will be tested for H. pylori infection. They will be randomly selected to represent the chosen population and invited to participate in the study based on informed consent. Confirmed infections will be treated by available combined therapy in line with treatment guidelines and the success of eradication will be retested during a control check-up.

Patients who will provide their consent to participate will undertake an interview about the risk factors in early childhood and their habits regarding alcohol consumption and use of tobacco. Compliance to testing and treatment, treatment results, adverse effects and reasons for dropping out will be additionally monitored. Gathered data will be analysed in alignment with our research questions. The investigators will disseminate reports and present the results to both the general public and the scientific community in order to foster future developments in gastric cancer prevention.

DETAILED DESCRIPTION:
The main objective of this study is to assess the feasibility of population-based H. pylori test-and-treat strategy for gastric cancer prevention in Europe. The study will allow to assess the feasibility of implementing H. pylori test-and-treat program in an early 30's age group at the population level, which will be carried out for the first time in Europe. This will come with scientifically valid assessment of programme processes, acceptance, effectiveness and possible adverse consequences.

The assessment of predefined quality indicators and achievements of each project task will consequently allow us to scale up the project to the national level, for example, by instituting a national program for gastric cancer prevention with population-based H. pylori test-and-treat program in the asymptomatic population around 30 years of age in different EU countries. The implementation of this strategy as a national program could result in significantly reduced gastric cancer incidence, disease burden and costs of other H. pylori-related diseases in the medium and long term in Slovenia and other participating countries, thus serving as a model for the implementation of this strategy in Europe.

The results of the study can help to guide other EU countries with intermediate and high gastric cancer incidence when implementing similar strategies. The results can also help to guide EU countries with low gastric cancer incidence when implementing similar programs for their subpopulations at risk (e.g. family members of patients with gastric cancer and immigrants from countries with high H. pylori infection and gastric cancer incidence). If implemented in a young adult population, the program can prevent further spread of H. pylori infection by curing the infection before or when they have just started their own families, therefore reducing the risk of intrafamilial transmission.

As shown in previously published economic evaluations of the strategy, the program is not only cost-effective in gastric cancer prevention but also in other high-risk areas. Besides that, H. pylori eradication will also prevent other serious clinical complications, such as peptic ulcers, dyspepsia, primary immune thrombocytopenia and anaemia caused by H. pylori infection.

In total, seven research centers from different European countries participate in the study - Croatia, Ireland, Latvia, Poland, Romania, and Slovenia. A predefined population of young people between 30 to 34 years of age will be invited to participate in the study. Based on signed informed consent they will be offered testing for H. pylori infection.

Acceptability and participation rate of the H. pylori test-and-treat strategy, the prevalence of H. pylori infection in the population of young adults, compliance with the 14-days treatment scheme, the eradication rate, and any adverse effects of the treatment in the population will be thoroughly assessed. Testing and treatment procedure will be substantiated with data about early childhood risk factors for H. pylori infection and the use of tobacco and alcohol consumption. Method used for capturing the participants' self-reported data will be a questionnaire administered by a health professional or self-administered by the patient.

Each center has its own specific research design:

1. Clinical Hospital Center Rijeka (KBC Rijeka), Croatia: 13C-urea breath test (UBT) confirmatory testing combined with H. pylori serology will be determined. H. pylori positive patients will be treated by bismuth-based quadruple therapy (Protocol I):

   • Protocol I with penicillin includes the following medications: Antibiotic 1 - Amoxicillin 4 x 500 mg or Clarithromycin 2 x 400 mg, Antibiotic 2 - Metronidazole 4 x 400 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg, Colloidal bismuth - Bismuth oxide 4 x 120 mg.

   In case there will be a treatment failure after Protocol I is completed, the remaining patients with a positive infection will be referred to a secondary treatment (Protocol II):

   • Protocol II includes the following medications: Antibiotic 1 - Levofloxacin 1 x 500 mg, Antibiotic 2 - Metronidazole 4 x 400 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg, Colloidal bismuth - Bismuth oxide 4 x 120 mg. All medications included in Protocol I or Protocol II will be taken orally for 14 consecutive days. After Protocol II is completed, the remaining patients with persisting infection will be treated by gastroenterologist according clinical practice guidelines.
2. University Hospital Centre Zagreb (KBC Zagreb), Croatia: 13C-urea breath test (UBT) confirmatory testing will be determined. In case of positive results participants will be treated with bismuth-based quadruple therapy (Protocol I). One month following the treatment a control UBT will be performed in order to confirm eradication. In case of treatment failure participants will be treated with second-line treatment (Protocol II).
3. Beacon Hospital, Ireland: H. pylori serology with high sensitivity will be offered to participants. For participants with positive serology test results, an additional UBT confirmatory testing will be the second step to confirm an active infection. H. pylori positive patients will be treated by bismuth-based quadruple therapy (Protocol I). One month after conclusion of the treatment a control UBT will be used to confirm eradication. Patients with treatment failure will be treated with an additional second protocol (Protocol II) according to local recommendations.
4. University of Latvia, Latvia: participants will be tested for H. pylori infection by UBT. H. pylori positive participants will be offered standard triple therapy for 14 days as the first-line therapy:

   Antibiotic 1 - Amoxicillin 2 x 1000 mg, Antibiotic 2 - Clarithromycin 2 x 500 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg.

   At least 30 days after the treatment participants will be retested for H. pylori by UBT to confirm eradication. Participants with treatment failure will be recommended second line treatment - levofloxacin-based:

   Antibiotic 1 - Levofloxacin 2 x 500 mg, Antibiotic 2 - Amoxicillin 2 x 1000 mg, Proton pump inhibitor - Esomeprazole 2 x 40 mg

   Or Pylera based:

   Antibiotic 1 - Metronidazole 4 x 125 mg Antibiotic 2 - Tetracycline 4 x 125 mg Colloidal bismuth - Bismuth Subcitrate Potassium 4 x 140 mg Proton pump inhibitor - Esomeprazole 2 x 40 mg
5. Uniwersytet medyczny we Wrocławiu, Poland: participants will be tested for H. pylori infection by locally validated H. pylori serology test. In case of a positive result the UBT will be performed for confirmation. Positive patients will be treated with bismuth-based quadruple therapy (Protocol I) followed by control UBT in order to confirm eradication. Treatment failure participants will be treated with second line treatment (Protocol II).
6. Iuliu Hațieganu University of Medicine and Pharmacy (UMF), Romania: Locally validated H. pylori serology with high sensitivity will be offered to participants. For participants with positive serology test results, additional UBT confirmatory testing will be the second step to confirm an active infection. H. pylori positive patients with be treated by bismuth-based quadruple therapy (Protocol I). One month after conclusion of the treatment a control UBT will be used to confirm eradication. Patients with treatment failure will be treated with additional second protocol (Protocol II) according to local recommendations.
7. National Institute of Public Health (NIJZ), Slovenia: Locally validated H. pylori serology with high sensitivity will be offered to participants. For participants with positive serology test results, additional UBT confirmatory testing will be the second step to confirm an active infection. H. pylori positive patients with be treated by bismuth-based quadruple therapy (Protocol I). One month after the conclusion of the treatment a control UBT will be used to confirm eradication. Patients with treatment failure will be treated with an additional second protocol (Protocol II) according to local recommendations.

The study will be conducted, commencing in 2024 and concluding in 2026. This timeframe has been chosen to allow for participant recruitment, conducting the study and data analysis for a thorough assessment of the feasibility of the proposed screening strategy.

ELIGIBILITY:
Inclusion Criteria:

* Young adults (generally 30 - 34 years of age)

Exclusion Criteria:

* Patients with mental or developmental limitations who cannot provide a fully-informed consent to participate (based on the assessment from research or patient's personal physician team)
* Previously treated H. pylori infection
* History of partial or total gastric resection due to benign or malign lesions

Ages: 30 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Infected adult patients by Helicobacter pylori
Sampling Method: Non-Probability Sample
Enrollment: 6800 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Healthcare workers' assessment of feasibility and acceptability of the proposed practical implementation of a screening program | 1 year
  Responses to qualitative questions and summary statistics from a post-enrollment questionnaire for healthcare workers involved into the implementation of the screening program.

SECONDARY OUTCOMES:
Eradication rate of infection with H. pylori | 1 year
  Subtraction of 1) participants who were subjected to treatment failure of the primary therapy regimen from 2) all participants with an active H. pylori infection who underwent the quadruple therapy regimen.
Description of the adverse events profile | 1 year
  Qualitative records of all self-reported (or physician-reported) adverse events during and after primary (or secondary) eradication therapy regimen. All non-serious or serious adverse event will be reported.
Participation rate of subjects selected for the program | 1 year
  a) completion of the enrollment process (points a)-d)); b) completion of the prospective study (points e)-h)).
  Subtraction of 1) study participants who:
  1. did not respond to an invitation,
  2. signed the informed consent form but were not included in the study due to exclusion criteria,
  3. declined to take a serology test,
  4. declined to take any of the UBTs as specified in the study protocol,
  5. had their therapy postponed due to maternity reasons,
  6. declined to be re-treated after the treatment failure of primary therapy,
  7. voluntarily withdrew at any time during their participation in the study,
  8. withdrew from the study within points a)-g) combined, from 2) all participants invited in the study.
  The participation rate is measured in frequencies and percentage points (%).

CONTACTS AND LOCATIONS:
Locations (7):
- Croatia (2):
  - University Hospital Centre Zagreb, Zagreb, City of Zagreb
  - Clinical Hospital Center Rijeka, Rijeka
- Beacon Hospital, Dublin, Ireland
- Clinical and Preventive Medicine of the University of Latvia, Riga, Latvia
- Wroclaw Medical University, Wroclaw, Poland
- Iuliu Hatieganu University of Medicine and Pharmacy, Cluj-Napoca, Cluj, Romania
- National Institute of Public Health, Slovenia, Ljubljana, Slovenia

REFERENCES:
- See also: Related Info — http://togas.lu.lv